CLINICAL TRIAL: NCT07333690
Title: The Effect of Healthy Lifestyle Management Education and Personalized Physical Activity Counseling on Pain, Functionality, Exercise Adherence, and Irisin Level in Patients With Knee Osteoarthritis: A Randomized Controlled Trial
Brief Title: The Effects of Healthy Lifestyle Management Training and Personalized Physical Activity Counseling: A Randomized Controlled Trial
Acronym: RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammed ARCA (Other)
Responsible Party: Sponsor-Investigator, Muhammed ARCA, Director, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Organization: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FZT-OA-Intervention-631
Record Dates: First submitted 2025-12-17; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Physical Activity; Exercise Therapy; Supervised Exercise; Randomized Controlled Trial
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physiotherapist-Supervised Intervention Group (Experimental): Participants will receive conventional physiotherapy combined with physiotherapist-supervised lifestyle management education and individualized physical activity counseling for 6 weeks, followed by a 6-week telephone-based follow-up.
  Interventions: Other: Physiotherapist-Supervised Intervention
- Home-Based Self-Managed Intervention Group (Active Comparator): Participants will receive lifestyle management education and an individualized home-based physical activity program, which they will perform independently without direct physiotherapist supervision.
  Interventions: Other: Physiotherapist-Supervised Intervention; Other: Home based self managed
- Control Group (Other): Participants will receive conventional physiotherapy only, as routinely applied in the hospital setting.
  Interventions: Other: Control

INTERVENTIONS:
Other: Physiotherapist-Supervised Intervention — Conventional Physiotherapy
  Lifestyle Management Education
  Individualized Physical Activity Counseling
  Arms: Home-Based Self-Managed Intervention Group; Physiotherapist-Supervised Intervention Group
Other: Home based self managed — Conventional Physiotherapy Lifestyle Management Education Individualized Physical Activity Counseling
  Arms: Home-Based Self-Managed Intervention Group
Other: Control — Conventional Physiotherapy
  Arms: Control Group

SUMMARY:
Knee osteoarthritis is a common condition that causes knee pain, stiffness, and difficulty in daily activities. Physical activity and exercise are recommended as part of the treatment; however, many individuals have difficulty maintaining regular exercise over time.

The purpose of this study is to evaluate the effects of different physical activity intervention approaches on pain, physical function, and exercise adherence in individuals with knee osteoarthritis. Participants will be randomly assigned to one of three groups. One group will receive a physiotherapist-supervised exercise and physical activity program. The second group will follow an individualized home-based physical activity program that they will perform independently after receiving initial instruction. The third group will receive usual care and will serve as the control group.

The intervention period will last six weeks. Participants in the intervention groups will then be followed for an additional six weeks using telephone-based follow-up to monitor adherence and ongoing physical activity. Outcomes related to pain, physical function, physical activity, and adherence to exercise will be assessed at different time points during the study.

The results of this study are expected to improve understanding of how supervised and home-based physical activity programs may contribute to the management of knee osteoarthritis and support the development of effective rehabilitation strategies.

DETAILED DESCRIPTION:
Knee osteoarthritis is a common musculoskeletal condition characterized by pain, reduced physical function, and limitations in daily activities. Regular physical activity and exercise are strongly recommended for the management of knee osteoarthritis; however, long-term adherence to exercise programs remains a major challenge for many patients.

The aim of this randomized controlled trial is to investigate the effects of different modes of physical activity intervention, in addition to usual care, on pain, physical function, exercise adherence, and selected cardiometabolic biomarkers in individuals with knee osteoarthritis.

Eligible participants diagnosed with knee osteoarthritis will be randomly allocated into one of three groups. The first group will receive a physiotherapist-supervised intervention, consisting of structured exercise sessions combined with personalized physical activity counseling delivered by a physiotherapist. The second group will receive an individualized home-based intervention, in which participants will perform the prescribed exercise and physical activity program independently at home following initial instruction and guidance. The third group will serve as the control group and will receive usual care only.

The intervention period will last six weeks for both intervention groups. Following the intervention phase, participants in the intervention groups will be followed for an additional six weeks through telephone-based monitoring to support adherence and record ongoing physical activity. Outcome assessments will be conducted at baseline, at the end of the six-week intervention period, and after completion of the follow-up period.

Primary outcomes will include pain intensity and physical function. Secondary outcomes will include exercise adherence, physical activity level, and selected cardiometabolic biomarkers. The results of this study are expected to provide evidence on the comparative effectiveness of supervised versus home-based physical activity interventions for individuals with knee osteoarthritis and to inform clinical practice and rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years

Diagnosed with knee osteoarthritis according to clinical and/or radiological criteria

Ability to walk independently

Willingness to participate and provide written informed consen

Exclusion Criteria:

* History of knee surgery within the last 6 months

Inflammatory rheumatic diseases

Neurological or cardiovascular conditions limiting physical activity

Participation in a structured exercise program within the last 3 months

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Physical Function | Baseline, Week 6, Week 12
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function subscale will be used to assess the physical functional status of the patients. This subscale consists of 17 items. Each item is scored on a Likert scale from 0 to 4 (0 = None, 4 = Extreme). The total score for this subscale ranges from 0 to 68 points, where higher scores indicate worse physical function (greater functional limitation).
Pain Severity | Baseline, Week 6, Week 12
  Numeric Analog Scale (NAS) Pain intensity will be assessed using the Numerical Rating Scale (NRS). The scale consists of a single item where patients rate their pain on a 11-point scale ranging from 0 to 10. A score of 0 represents "no pain" and a score of 10 represents "the worst possible pain." Higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
Exercise Adherence Rating Scale | Baseline, Week 6, Week 12
  The Exercise Adherence Rating Scale (EARS) will be used to measure the patients' adherence to the prescribed exercise program. The scale (Section B) consists of 6 items. Each item is scored on a 5-point Likert scale (0 = Completely Agree, 4 = Completely Disagree). The total score ranges from 0 to 24, where higher scores indicate better adherence to the exercise program.
Serum Irisin Level | Baseline, Week 6, Week 12
  Serum irisin concentrations will be measured using an Enzyme-Linked Immunosorbent Assay (ELISA) kit.

IPD SHARING:
Plan to Share IPD: No
In accordance with the personal data privacy law, information will not be shared with third parties.